CLINICAL TRIAL: NCT00691171
Title: Using an Electronic Health Record-based Intervention and Broad Education Reach Strategies to Improve Quality of Care for GERD and Gastroprotection for Patients on NSAIDs: a Randomized Controlled Trial
Brief Title: Electronic Health Record (EHR)-Based Intervention for Gastroesophageal Reflux Disease (GERD) and Chronic Non-steroidal Anti-inflammatory Drug (NSAID) Use
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GUS-DUM-2007/1
Record Dates: First submitted 2008-05-30; First posted 2008-06-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: GERD
Keywords: gastroesophageal reflux disease; GERD; nonsteroidal anti-inflammatory drugs; peptic ulcer; Diagnosed GERD; Atypical GERD symptoms; chronic NSAID therapy; Risk for ulcer
MeSH Terms: conditions — Gastroesophageal Reflux; Peptic Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: GERD: Patients with established diagnoses of GERD based on ICD-9 codes
- 2: Atypical GERD: Patients without an established diagnosis of GERD with atypical symptoms that could be due to GERD (e.g., asthma)
- 3: Chronic NSAID users: Patients using chronic NSAIDs who are at increased risk of GI complications (defined as previous diagnosis of peptic ulcer disease; age 75 or older; or concomitant use of corticosteroids, anticoagulants, or aspirin)

SUMMARY:
The purpose of the study is to examine the impact of augmented, high-quality physician-coordinated care executed via an electronic health record (EHR)-based intervention on quality of care for gastroesophageal reflux disease (GERD) and for gastroprotection for patients on chronic non-steroidal anti-inflammatory drugs (NSAIDs) at increased risk for upper GI tract ulcers and ulcer related complications.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility as determined by criteria for participation in studies as part of the MQIC
* Agreement of participating clinical practices to undergo training in the electronic health record (EHR) intervention designed for this study

Exclusion Criteria:

* Based on voluntary participation by MQIC practices, so practices were excluded if they decided to opt out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primarily primary care practices of physicians participating in the Medical Quality Improvement Consortium (MQIC)
Sampling Method: Non-Probability Sample
Enrollment: 5234 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Diagnoses of GERD | After 12 months of intervention
Prescriptions for gastroprotective medicines in at-risk, chronic NSAID users | After 12 months of intervention

SECONDARY OUTCOMES:
Prescriptions for GERD medications | After 12 months of intervention
Change in GERD symptoms score | After 12 months of intervention
NSAID-related GI complications | After 12 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: James M Gill, MD, PhD, Principal Investigator — Delaware Valley Outcomes Research

REFERENCES:
- [Result] Gill JM, Mainous AG 3rd, Koopman RJ, Player MS, Everett CJ, Chen YX, Diamond JJ, Lieberman MI. Impact of EHR-based clinical decision support on adherence to guidelines for patients on NSAIDs: a randomized controlled trial. Ann Fam Med. 2011 Jan-Feb;9(1):22-30. doi: 10.1370/afm.1172. PMID 21242557